CLINICAL TRIAL: NCT06620536
Title: Restoring Hand Function in Patients with Tetraplegia by Intraneural Stimulation of Peripheral Nerves
Acronym: REGRASP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGRASP
Record Dates: First submitted 2024-09-13; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Tetraplegics
Keywords: electrodes; intraneural stimulation; hand; tetraplegia
MeSH Terms: conditions — Quadriplegia | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Restoring hand function in patients with tetraplegia by intraneural stimulation of peripheral nerves (Experimental)
  Interventions: Device: Electrical stimulation

INTERVENTIONS:
Device: Electrical stimulation — Electrical stimulation of peripheral nerves for the recovery of hand function in tetraplegic patients of fundamental importance in improving quality of life.

SUMMARY:
The aim of the clinical investigation is to evaluate the feasibility, in terms of efficacy and safety, of a prosthetic system, the Regrasp 1 system, based on intraneural stimulation via TIME- 4H electrodes, as an aid device for restoring hand function in tetraplegic patients.

DETAILED DESCRIPTION:
The study involves implanting intraneural electrodes in the nerve used to open and close the hand.

Electrical stimulation will activate the forearm and hand muscles, and thus evoke movements such as opening and closing the fingers of the hand and wrist movements. Electrodes will be implanted temporarily and reversibly within the fascicles so that a more selective and therefore more effective stimulation can be determined. The electrodes will remain implanted for about 6 months.

During this period, the results of the external electrical stimulation will be analysed through experimental sessions that will take place at the Careggi University Hospital. At the end of the study, the electrodes will be removed by surgery under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged between 18 and 70.
2. Spinal cord injury at the C5-6 level, with complete motor paralysis (ASIA A or ASIA B).
3. Chronic injury (> 6 months), with stable clinical condition.

Exclusion Criteria:

1. Systemic infections.
2. Central and/or peripheral nervous system comorbidity.
3. Reduced joint flexibility.
4. Severe spasticity of the upper limb (mAS 3).
5. Severe denervation of forearm and hand muscles (as demonstrated by electromyography and electroneurography analysis and intraoperative neural stimulation).
6. Muscles not electrically excitable.
7. Presence of hyperalgesia or allodynia.
8. Wearers of life support devices that could be adversely affected by electromagnetic interference, such as pacemakers, implanted cardioverter defibrillators, etc.
9. Cognitive impairment.
10. Active or history of psychiatric illnesses including major depression, bipolar disorder and personality disorders (borderline or antisocial personality disorder).
11. Pregnancy.
12. History of alcohol or substance abuse.
13. Acquired brain injury with residual deficits.
14. Participation in other clinical trials.
15. Known allergies/hypersensitivity to TIME-4H electrode materials.
16. Life expectancy of less than one year.
17. Contraindications to general anaesthesia (patient refusal, severe aortic stenosis, significant pulmonary disease, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of REGRASP device, regarding muscle selectivity | from baseline to follow-up at month 6
  The muscle selectivity index will be obtained by intraneural stimulation with a TIME-4H astimulator. Single stimulation pulses (1 Hz) will be applied from each active site of each implanted TIME-4H electrode. Simultaneously, electromyographic (EMG) signals of the flexor and extensor muscles of the forearm and hand, innervated by the median and radial nerves, respectively, will be recorded. For the EMG acquisitions we will use the CE-marked Sessantaquattro+ system. The peak-to-peak value of the compound muscle action potential (CMAP), evoked by each stimulation pulse, will be calculated and normalised with respect to the maximum value obtained for each muscle during the overall experimental session. These normalised levels of muscle activation will be used to define the relationship between current intensity and muscle recruitment for each active site and so to calculate an index of muscle selectivity.
efficacy of REGRASP device, regarding muscle functional selectivity | from baseline to follow-up at month 6
  To assess functional selectivity, bursts of stimulation, with a duration of 0.5-1 sec, will be applied from each active site of each implanted TIME-4H. Evoked movements will be assessed using the Medical Research Council (MRC) scale. In addition, we will characterise evoked movements in terms of muscle activity patterns by recording the EMG activity of the muscles with the Sessantaquattro+ system, and in terms of kinematic patterns (amplitude and velocity) and generated force. The same experiments will then be performed by modulating the frequency of the stimulation bursts (in the range 10-100 Hz) while keeping the amplitude fixed at a value capable of generating functional movements. Thus, we will evaluate the possibility of gradually controlling the amplitude and force of the movement by adjusting the different stimulation parameters.
Muscle fatigue | from baseline to follow-up at month 6
  To measure muscle fatigue, experiments will be conducted in which stimulation trains will be applied for approximately 20-30 seconds. At the same time, the EMG activity of the forearm and hand muscles and the grip force generated will be recorded. Some indices of muscle fatigue found in the literature will then be calculated, which measure, for example, the rate at which muscle strength decreases over time. The values obtained will be compared with those measured during voluntary contractions and with those induced by other stimulation modalities, such as FES with surface electrodes.
Functional recovery analysis | from baseline to follow-up at month 6
  Restoration of hand function, in particular grasping movements and manipulation of objects, when the patient is assisted by the neuroprosthetic system. This will be assessed using four different tests with related score:
  * the Grasp and Release test, awarded on the basis of the number of objects the patient is able to manipulate and the number of repetitions they are able to perform in a specific time interval;
  * ADL test, used to evaluate the performance of the neuroprosthetic system when used during activities of daily living;
  * GRASSP, a measure of clinical impairment that incorporates three vital domains of upper limb function: sensation, strength and grip;
  * SCIM, a disability scale developed to specifically assess the ability of spinal cord injury patients to perform basic activities of daily living independently.

SECONDARY OUTCOMES:
to evaluate possible plastic changes in the central nervous system induced by the use of the neuroprosthetic system. | from baseline to follow-up at month 6
  Somatosensory cortical mapping of the paralysed hand will be performed using somatosensory evoked potentials (PESs). The median and ulnar nerves will be stimulated using bipolar surface electrodes at a frequency of 1 Hz. The amplitude of the response will be measured automatically by the BE Plus PRO system, as the difference between the peak potential and the signal baseline, for each electrode.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy, Italy